CLINICAL TRIAL: NCT02792231
Title: A Randomized, Double-blind, Double-dummy, Parallel-group Study Comparing the Efficacy and Safety of Ofatumumab Versus Teriflunomide in Patients With Relapsing Multiple Sclerosis.
Brief Title: Efficacy and Safety of Ofatumumab Compared to Teriflunomide in Patients With Relapsing Multiple Sclerosis.
Acronym: ASCLEPIOS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMB157G2302; 2015-005419-33 (EudraCT Number)
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Relapsing Multiple Scelrosis
Keywords: Relapsing multiple sclerosis; Ofatumumab; adult; OMB157; multiple sclerosis; T1 lesions; T2 lesions; relapse; GD-enhancing MRI; McDonald criteria; RRMS; SPMS
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OMG 20 mg (Experimental): Ofatumumab 20 mg pre-filled syringes for subcutaneous injectionon on days 1
  ,7 ,14, week 4 and every 4 weeks thereafter and a teriflunomide-matching placebo, taken orally once daily
  Interventions: Drug: Ofatumumab subcutaneous injection; Drug: Teriflunomide-matching placebo capsules
- TER 14 mg (Active Comparator): Teriflunomide 14 mg oral capsule taken once daily and matching placebo for subcutaneous injections to ofatumumab on days 1, 7, 14, week 4 and every 4 weeks thereafter
  Interventions: Drug: Teriflunomide capsule; Drug: Matching placebo of ofatumumab subcutaneous injections

INTERVENTIONS:
Drug: Ofatumumab subcutaneous injection — Ofatumumab 20 mg prefilled syringes for subcutaneous injection on days 1, 7, 14, week 4 and every 4 weeks thereafter
  Arms: OMG 20 mg
Drug: Teriflunomide-matching placebo capsules — Placebo capsule, matching in appearance to teriflunomide, taken orally once daily
  Arms: OMG 20 mg
Drug: Teriflunomide capsule — Teriflunomide 14 mg oral capsule taken once daily
  Arms: TER 14 mg
Drug: Matching placebo of ofatumumab subcutaneous injections — Matching placebo of ofatumumab subcutaneous injections on days 1, 7, 14, week 4 and every 4 weeks thereafter
  Arms: TER 14 mg

SUMMARY:
To compare the efficacy and safety of ofatumumab administered subcutaneously (sc) every 4 weeks versus teriflunomide administered orally once daily in patients with relapsing multiple sclerosis

DETAILED DESCRIPTION:
This was a randomized, double-blind, double-dummy, active comparatorcontrolled, parallel-group, multi-center study with variable treatment duration in approximately 900 patients with relapsing multiple sclorosis (RMS). The maximal treatment duration in the study for an individual patient was 2.5 years. Eligible patients were randomized to receive either experimental ofatumumab subcutaneous (s.c.) injections every 4 weeks or active comparator teriflunomide orally once daily. The dose regimen for ofatumumab for this study was a loading dose regimen of 20 mg at Day 1, Day 7 and Day 14, followed by a maintenance dose regimen of 20 mg administered every 4 weeks starting at Week 4. In order to blind for the different formulations, double-dummy masking was used, i.e., all patients will take injections (containing either active ofatumumab or placebo) and oral capsules (containing either active teriflunomide or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 55 years at Screening
* Diagnosis of multiple sclerosis (MS)
* Relapsing MS: relapsing-remitting MS (RRMS) or secondary progressive MS (SPMS) with disease activity
* Documentation of at least: 1 relapse during the previous 1 year OR 2 relapses during the previous 2 years OR a positive gadolinium-enhancing MRI scan during the year prior to randomization
* Disability status at Screening with an Expanded Disability Status Scale (EDSS) score of 0 to 5.5
* Neurologically stable within 1 month prior to randomization

Exclusion Criteria:

* Patients with primary progressive MS or SPMS without disease activity
* Disease duration of more than 10 years in patients with an EDSS score of 2 or less
* Patients with an active chronic disease of the immune system other than MS
* Patients at risk of developing or having reactivation of hepatitis
* Patients with active systemic infections or with neurological findings consistent with PML

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 955 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis
Locations (160):
- United States (54):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Cullman, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Basalt, Colorado
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Centennial, Colorado
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Fairfield, Connecticut
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Oldsmar, Florida
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Palm Coast, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Suwanee, Georgia
  - Novartis Investigative Site, Anderson, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Wellesley, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Golden Valley, Minnesota
  - Novartis Investigative Site, Billings, Montana
  - Novartis Investigative Site, Great Falls, Montana
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Westerville, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Willow Grove, Pennsylvania
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Cordova, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Greenville, Texas
  - Novartis Investigative Site, Lubbock, Texas
  - Novartis Investigative Site, Sherman, Texas
  - Novartis Investigative Site, Orem, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Kirkland, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Waukesha, Wisconsin
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán
- Novartis Investigative Site, Liverpool, New South Wales, Australia
- Novartis Investigative Site, Vienna, Austria
- Belgium (4):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (4):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
- Croatia (2):
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Zagreb
- Czechia (5):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Havířov, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Ostrava-Poruba
  - Novartis Investigative Site, Prague
- Finland (2):
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (7):
  - Novartis Investigative Site, Nice, Cedex1
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
- Germany (13):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
- Hungary (2):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Esztergom, HUN
- India (6):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Mumbai
- Italy (6):
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Rome
- Latvia (2):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Riga
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Novartis Investigative Site, Chihuahua City, Mexico
- Novartis Investigative Site, Drammen, Norway
- Peru (3):
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, Lima
- Poland (5):
  - Novartis Investigative Site, Głogów
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zabrze
- Portugal (8):
  - Novartis Investigative Site, Matosinhos Municipality, Porto District
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Loures
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Santa Maria da Feira
- Russia (7):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (3):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Ružomberok
- South Africa (2):
  - Novartis Investigative Site, Pretoria
  - Novartis Investigative Site, Rosebank
- Spain (6):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Lugano, Switzerland
- Novartis Investigative Site, Tainan, Taiwan
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Haseki / Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Trabzon
- United Kingdom (3):
  - Novartis Investigative Site, Luton, Beds
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Williams MJ, Amezcua L, Cohan SL, Cohen JA, Delgado SR, Hua LH, Lucassen EB, Piccolo RS, Koulouris CR, Stankiewicz J. Efficacy of Ofatumumab and Teriflunomide in Patients With Relapsing MS From Racial/Ethnic Minority Groups: ASCLEPIOS I/II Subgroup Analyses. Neurology. 2024 Aug 13;103(3):e209610. doi: 10.1212/WNL.0000000000209610. Epub 2024 Jul 17. PMID 39018512
- [Derived] Bhan V, Clift F, Baharnoori M, Thomas K, Patel BP, Blanchette F, Adlard N, Vudumula U, Gudala K, Dutta N, Grima D, Mouallif S, Farhane F. Cost-consequence analysis of ofatumumab for the treatment of relapsing-remitting multiple sclerosis in Canada. J Comp Eff Res. 2023 Sep;12(9):e220175. doi: 10.57264/cer-2022-0175. Epub 2023 Aug 22. PMID 37606897
- [Derived] Gartner J, Hauser SL, Bar-Or A, Montalban X, Cohen JA, Cross AH, Deiva K, Ganjgahi H, Haring DA, Li B, Pingili R, Ramanathan K, Su W, Willi R, Kieseier B, Kappos L. Efficacy and safety of ofatumumab in recently diagnosed, treatment-naive patients with multiple sclerosis: Results from ASCLEPIOS I and II. Mult Scler. 2022 Sep;28(10):1562-1575. doi: 10.1177/13524585221078825. Epub 2022 Mar 10. PMID 35266417
- [Derived] Hauser SL, Bar-Or A, Cohen JA, Comi G, Correale J, Coyle PK, Cross AH, de Seze J, Leppert D, Montalban X, Selmaj K, Wiendl H, Kerloeguen C, Willi R, Li B, Kakarieka A, Tomic D, Goodyear A, Pingili R, Haring DA, Ramanathan K, Merschhemke M, Kappos L; ASCLEPIOS I and ASCLEPIOS II Trial Groups. Ofatumumab versus Teriflunomide in Multiple Sclerosis. N Engl J Med. 2020 Aug 6;383(6):546-557. doi: 10.1056/NEJMoa1917246. PMID 32757523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was pre-specified in the protocol to combine the data from this study with study NCT02792218 (COMB157G2301) for some outcome measures. Please refer to NCT02792218 for Participant Flow information for participants from other study.
Pre-assignment Details: A total of 1280 patients were screened, of whom 955 patients were randomized into the study.
Groups:
- OMB 20 mg: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter (+ teriflunomide-matching placebo capsule orally once daily)
- TER 14 mg: Teriflunomide 14 mg capsule orally once daily (+ ofatumumab-matching placebo injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter)
Period: Overall Study
Arm/Group | OMB 20 mg | TER 14 mg
Started | 481 | 474
Completed | 399 | 390
Not Completed | 82 | 84
Not completed — Patient/guardian decision | 32 | 42
Not completed — Adverse Event | 15 | 11
Not completed — Physician Decision | 14 | 12
Not completed — Lack of Efficacy | 7 | 9
Not completed — Lost to Follow-up | 9 | 5
Not completed — Pregnancy | 1 | 3
Not completed — Non-compliance with study treatment | 2 | 1
Not completed — Protocol deviation | 2 | 0
Not completed — Technical problems | 0 | 1

BASELINE CHARACTERISTICS:
Population: It was pre-specified in the protocol to combine the data from this study with study NCT02792218 (COMB157G2301) for some outcome measures. Please refer to NCT02792218 for Baseline information for participants from other study.
Groups:
- Total: Total of all reporting groups
Arm/Group | OMB 20 mg | TER 14 mg | Total
Number analyzed (Participants) | 481 | 474 | 955
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (9.28) | 38.2 (9.47) | 38.1 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319 | 319 | 638
  Male | 162 | 155 | 317
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 21 | 19 | 40
  Black or African American | 13 | 18 | 31
  White | 418 | 417 | 835
  Other | 20 | 14 | 34
  Unknown | 9 | 6 | 15
Number of relapses in the past 12 months prior to screening [Mean (Standard Deviation); unit: Number of relapses] — Reported numbers are from investigator records
  Number of relapses | 1.3 (0.74) | 1.3 (0.73) | 1.3 (0.74)
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: Score on a scale] — The EDSS uses an ordinal scale to assess neurologic impairment in MS based on a neurological examination. Scores in each of 7 functional systems (Visual, Brain Stem, Pyramidal, Cerebellar,Sensory, Bowel & Bladder, and Cerebral) and an ambulation score were combined to determine the EDSS steps, ranging from 0 (normal) to 10 (death due to MS). Population: Participants with data that met requirements for analysis were included
  Score on a scale
    number analyzed (Participants) | 481 | 473 | 954
    (all) | 2.90 (1.343) | 2.86 (1.373) | 2.88 (1.358)
Number of gadolinium-enhancing T1 lesions [Mean (Standard Deviation); unit: T1 lesions] — Magnetic Resonance Imaging (MRI) scans of the brain were were read by the central MRI reading center. The central reading center was blinded with no access to information on treatment assignments Population: Participants with data that met requirements for analysis were included
  T1 lesions
    number analyzed (Participants) | 469 | 470 | 939
    (all) | 1.6 (4.07) | 1.5 (4.07) | 1.5 (4.07)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR)
Description: ARR was the number of confirmed relapses in a year, calculated as the total number of relapses for all participants in the treatment group divided by the total participant-years of time in study. A confirmed MS relapse was defined as one accompanied by a clinically-relevant change in the EDSS performed by the Independent EDSS rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores or 2 points on one functional score (excluding changes involving bowel/bladder or cerebral functional system). Comparisons were made to the previous rating (the last EDSS rating that did not occur during a relapse).
Time Frame: Baseline up to 2.5 years
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: number of relapses in a year
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 469 | 470
number of relapses in a year | 0.10 [0.08 to 0.13] | 0.25 [0.21 to 0.30]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; Obtained from fitting a negative binomial regression model with log-link to the number of relapses, adjusted for treatment and region as factors, number of relapses in previous year, baseline EDSS, baseline number of Gd-enhancing lesions and the patient's age at baseline as covariates. The natural log of the time-in-study was used as offset to annualize the relapse rate; Test type: Superiority; p < 0.001, negative binomial regression model; rate ratio = 0.416, 95% CI 2-sided [0.309 to 0.560]

2. Secondary Outcome: 3-month Confirmed Disability Worsening (3mCDW) Based on EDSS - Pooled Data
Description: A 3-month confirmed disability worsening (3mCDW) was defined as an increase from baseline in Expanded Disability Status Scale (EDSS) score sustained for at least 3 months. For patients with a baseline EDSS of 0, the criterion for disability worsening was an increase in EDSS of ≥1.5, for patients with a baseline EDSS of 1 to 5 or ≥5.5, the criterion for disability worsening was an increase in EDSS of ≥1 or ≥0.5, respectively. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint.
Time Frame: Baseline, every 3 months up to 2.5 years
Population: Full analysis set from combined studies
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 944 | 932
percentage of participants
  Month 18 - from Kaplan Meier estimates | 9.4 [7.6 to 11.5] | 13.5 [11.4 to 16.0]
  Month 24 - from Kaplan Meier estimates | 10.9 [8.8 to 13.4] | 15.0 [12.6 to 17.7]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; Pooled data - this study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint; Test type: Superiority; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 0.657, 95% CI 2-sided [0.500 to 0.863]

3. Secondary Outcome: 3-month Confirmed Disability Worsening (3mCDW) Based on EDSS - Study COMB157G2302
Description: as for outcome 2
Time Frame: Baseline, every 3 months up to 2.5 years
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 479 | 473
percentage of participants
  Month 18 - from Kaplan Meier estimates | 9.3 [6.9 to 12.5] | 13.2 [10.3 to 16.7]
  Month 24 - from Kaplan Meier estimates | 10.5 [7.8 to 14.1] | 14.6 [11.5 to 18.6]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint; Test type: Superiority; p = 0.038, Regression, Cox; Hazard Ratio (HR) = 0.662, 95% CI 2-sided [0.449 to 0.977]

4. Secondary Outcome: 6-month Confirmed Disability Worsening (6mCDW) Based on EDSS - Pooled Data
Description: A 6-month confirmed disability worsening (6mCDW) was defined as an increase from baseline in Expanded Disability Status Scale (EDSS) score sustained for at least 6 months. For patients with a baseline EDSS of 0, the criterion for disability worsening was an increase in EDSS of ≥1.5, for patients with a baseline EDSS of 1 to 5 or ≥5.5, the criterion for disability worsening was an increase in EDSS of ≥1 or ≥0.5, respectively. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint.
Time Frame: Baseline, every 3 months up to 2.5 years
Population: Full analysis set from combined studies
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 944 | 932
percentage of participants
  Month 18- from Kaplan Meier estimates | 7.8 [6.2 to 9.7] | 10.7 [8.9 to 13.0]
  Month 24 - from Kaplan Meier estimates | 8.1 [6.5 to 10.2] | 12.0 [9.9 to 14.5]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.012, Regression, Cox; Hazard Ratio (HR) = 0.676, 95% CI 2-sided [0.498 to 0.917]

5. Secondary Outcome: 6-month Confirmed Disability Worsening (6mCDW) Based on EDSS - Study COMB157G2302
Description: as for outcome 4
Time Frame: Baseline, every 3 months up to 2.5 years
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 479 | 473
percentage of participants
  Month 18- from Kaplan Meier estimates | 8.0 [5.9 to 11.0] | 10.0 [7.5 to 13.2]
  Month 24 - from Kaplan Meier estimates | 8.0 [5.9 to 11.0] | 10.9 [8.2 to 14.4]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.215, Regression, Cox; Hazard Ratio (HR) = 0.759, 95% CI 2-sided [0.490 to 1.174]

6. Secondary Outcome: 6-month Confirmed Disability Improvement (6mCDI ) Based on EDSS - Pooled Data
Description: A 6-month confirmed disability improvement (6mCDI) was defined as a decrease from baseline EDSS sustained for at least 6 months. For patients with a baseline EDSS of 0 to 1.5, no disability improvement was possible based on the protocol definition of an improvement; for patients with a baseline EDSS of ≥2 to 6 or ≥6.5 to 9.5, the criterion for disability improvement was a decrease in EDSS of ≤1 or ≤0.5, respectively. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint.
Time Frame: Baseline, every 3 months up to 2.5 years
Population: Full analysis set from combined studies
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 749 | 724
percentage of participants
  Month 18 - from Kaplan Meier estimates: number analyzed (Participants) | 749 | 723
  Month 18 - from Kaplan Meier estimates | 10.1 [8.1 to 12.6] | 7.6 [5.8 to 9.8]
  Month 24 - from Kaplan Meier estimates: number analyzed (Participants) | 749 | 723
  Month 24 - from Kaplan Meier estimates | 11.0 [8.8 to 13.7] | 8.2 [6.3 to 10.6]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.092, Regression, Cox; Hazard Ratio (HR) = 1.355, 95% CI 2-sided [0.952 to 1.928]

7. Secondary Outcome: 6-month Confirmed Disability Improvement (6mCDI ) Based on EDSS - Study COMB157G2302
Description: as for outcome 6
Time Frame: Baseline, every 3 months up to 2.5 years
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 374 | 361
percentage of participants
  Month 18 - from Kaplan Meier estimates | 11.1 [8.2 to 14.8] | 8.1 [5.6 to 11.6]
  Month 24 - from Kaplan Meier estimates | 12.3 [9.1 to 16.5] | 8.1 [5.6 to 11.6]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.090, Regression, Cox; Hazard Ratio (HR) = 1.523, 95% CI 2-sided [0.936 to 2.477]

8. Secondary Outcome: Number of Gadolinium-enhancing T1 Lesions Per MRI Scan
Description: Total number of Gd-enhancing T1 lesions across all scans per patient adjusted for different number of scans due to variable follow-up time in study.
Time Frame: Baseline, yearly up to 2.5 years
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: lesions per scan
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 438 | 433
lesions per scan | 0.0317 [0.021 to 0.048] | 0.5172 [0.404 to 0.662]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; Test type: Superiority; p < .001, negative binomial regression model; rate ratio = 0.061, 95% CI 2-sided [0.037 to 0.101]

9. Secondary Outcome: Number of New or Enlarging T2 Lesions on MRI Per Year (Annualized Lesion Rate)
Description: Number of new/enlarging T2 lesions on last available MRI scan compared to baseline adjusted for different time of scans versus baseline due to variable follow up time in study
Time Frame: Baseline, yearly up to 2.5 years
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: T2 lesions per year
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 448 | 442
T2 lesions per year
  Month 12 n=422,410: number analyzed (Participants) | 422 | 410
  Month 12 n=422,410 | 0.94 [0.80 to 1.11] | 4.41 [3.83 to 5.08]
  Month 24 n=90,76: number analyzed (Participants) | 90 | 76
  Month 24 n=90,76 | 0.72 [0.51 to 1.02] | 3.72 [2.68 to 5.18]
  EOS n=448,442 | 0.64 [0.55 to 0.75] | 4.16 [3.64 to 4.75]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; Month 12; Test type: Superiority; p < .001, negative binomial regression model; rate ratio = 0.21, 95% CI 2-sided [0.17 to 0.27]
Statistical Analysis 2: Comparison: OMB 20 mg vs TER 14 mg; Month 24; Test type: Superiority; p < .001, negative binomial regression model; rate ratio = 0.19, 95% CI 2-sided [0.12 to 0.31]
Statistical Analysis 3: Comparison: OMB 20 mg vs TER 14 mg; End of Study; Test type: Superiority; p < .001, negative binomial regression model; rate ratio = 0.15, 95% CI 2-sided [0.13 to 0.19]

10. Secondary Outcome: Neurofilament Light Chain (NfL) Concentration in Serum
Description: The NfL concentration (geometric mean concentration) was estimated by treatment and time point with using a repeated measures model on the basis of all evaluable log-transformed NfL values.
Time Frame: Month 3, 12 and 24
Population: Full analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 425 | 423
pg/mL
  Month 3 n=425,423 | 8.92 [8.62 to 9.23] | 10.02 [9.68 to 10.36]
  Month 12 n=406,406: number analyzed (Participants) | 406 | 406
  Month 12 n=406,406 | 7.06 [6.77 to 7.37] | 9.53 [9.13 to 9.95]
  Month 24 n=345,349: number analyzed (Participants) | 345 | 349
  Month 24 n=345,349 | 6.80 [6.47 to 7.13] | 8.99 [8.57 to 9.44]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; Month 3; Test type: Superiority; p < .001, Mixed Models Analysis; Mixed Models for Repeated Measures (MMRM); Geo-mean ratio = 0.89, 95% CI 2-sided [0.85 to 0.93]
Statistical Analysis 2: Comparison: OMB 20 mg vs TER 14 mg; Month 12; Test type: Superiority; p < .001, Mixed Models Analysis; Mixed Models for Repeated Measures (MMRM); Geo-mean ratio = 0.74, 95% CI 2-sided [0.70 to 0.79]
Statistical Analysis 3: Comparison: OMB 20 mg vs TER 14 mg; Month 24; Test type: Superiority; p < .001, Mixed Models Analysis; Mixed Models for Repeated Measures (MMRM); Geo-mean ratio = 0.76, 95% CI 2-sided [0.71 to 0.81]

11. Secondary Outcome: Annualized Rate of Brain Volume Loss Based on Assessments of Percent Brain Volume Change From Baseline
Description: Percent change from baseline in brain volume loss (BVL) on all MRI scans adjusted for different time of scan versus baseline due to variable follow up time in study
Time Frame: Baseline, Months 12 and 24
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: percentage of brain volume loss
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 437 | 433
percentage of brain volume loss | -0.29 [-0.35 to -0.23] | -0.35 [-0.42 to -0.29]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; Test type: Superiority; p = 0.128, random coefficient model; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.02 to 0.15]

12. Secondary Outcome: Participants With Confirmed Relapse
Description: A confirmed MS relapse was defined as one accompanied by a clinically-relevant change in the EDSS performed by the Independent EDSS rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores or 2 points on one functional score (excluding changes involving bowel/bladder or cerebral functional system).
Time Frame: Baseline up to 2.5 years
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 469 | 470
percentage of participants | 16.51 [13.18 to 20.57] | 32.68 [28.10 to 37.79]

13. Secondary Outcome: Annualized Relapse Rate (ARR) >8 Weeks After Onset of Treatment
Description: as for outcome 1
Time Frame: Baseline up to 2.5 years
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: number of relapses in a year
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 461 | 467
number of relapses in a year | 0.096 [0.05 to 0.14] | 0.241 [0.16 to 0.32]

14. Secondary Outcome: 3-month Confirmed Disability Worsening (3mCDW) Based on EDSS > 8 Weeks After Onset of Treatment - Pooled Data
Description: as for outcome 2
Time Frame: Baseline up to 2.5 years
Population: Full analysis set from combined studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 944 | 932
percentage of participants
  Month 18 - from Kaplan Meier estimates | 9.4 [7.6 to 11.5] | 13.5 [11.4 to 16.0]
  Month 24 - from Kaplan Meier estimates | 10.9 [8.8 to 13.4] | 15.0 [12.6 to 17.7]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.641, 95% CI 2-sided [0.486 to 0.847]

15. Secondary Outcome: 6-month Confirmed Disability Worsening (6mCDW) Based on EDSS > 8 Weeks After Onset of Treatment - Pooled Data
Description: as for outcome 4
Time Frame: Baseline up to 2.5 years
Population: Full analysis set from combined studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 944 | 932
percentage of participants
  Month 18- from Kaplan Meier estimates | 7.8 [6.2 to 9.7] | 10.7 [8.9 to 13.0]
  Month 24 - from Kaplan Meier estimates | 8.1 [6.5 to 10.2] | 12.0 [9.9 to 14.5]
Statistical Analysis 1: Comparison: OMB 20 mg vs TER 14 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.008, Regression, Cox; Hazard Ratio (HR) = 0.657, 95% CI 2-sided [0.481 to 0.898]

16. Secondary Outcome: 6-month Confirmed Cognitive Decline on Symbol Digit Modalities Test (SDMT) - Pooled Data
Description: A 6-month confirmed cognitive decline was defined as a decrease from baseline of at least 4 points in SDMT score sustained for at least 6 months. Processing speed was measured by the Symbol Digit Modalities Test (SDMT) score. SDMT measures the time to pair abstract symbols with specific numbers. The test requires visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items in 90 seconds. (max=110, min=0). Higher scores indicate improvement. Lower scores indicate worsening. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint
Time Frame: Baseline, every 6 months up to 2.5 years
Population: Full analysis set from combined studies
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 930 | 917
percentage of participants
  Month 18 - from Kaplan Meier estimates | 14.3 [12.2 to 16.8] | 13.7 [11.5 to 16.1]
  Month 24 - from Kaplan Meier estimates | 15.4 [13.1 to 18.2] | 14.0 [11.8 to 16.6]

17. Secondary Outcome: 6-month Confirmed Disability Worsening (6mCDW) or 6-month Confirmed Cognitive Decline (6mCCD) - Pooled Data
Description: A 6-month confirmed disability worsening (6mCDW) was defined as an increase from baseline in Expanded Disability Status Scale (EDSS) score sustained for at least 6 months. For patients with a baseline EDSS of 0, the criterion for disability worsening was an increase in EDSS of ≥1.5, for patients with a baseline EDSS of 1 to 5 or ≥5.5, the criterion for disability worsening was an increase in EDSS of ≥1 or ≥0.5, respectively. A 6-month confirmed cognitive decline (6mCCD) was defined as a 4-point worsening on Symbol Digit Modalities Test (SDMT) sustained for at least 6 months. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint.
Time Frame: Baseline up to 2.5 years
Population: Full analysis set from combined studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 941 | 930
percentage of participants
  Month 18 - from Kaplan Meier estimates | 20.5 [18.0 to 23.4] | 21.7 [19.1 to 24.6]
  Month 24 - from Kaplan Meier estimates | 21.4 [18.8 to 24.3] | 22.6 [19.9 to 25.7]

18. Secondary Outcome: Change in Cognitive Performance Measured by the Symbol Digit Modalities Test (SDMT) - Pooled Data
Description: Processing speed is being measured by the Symbol Digit Modalities Test (SDMT) score. SDMT measures the time to pair abstract symbols with specific numbers. The test requires visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items in 90 seconds. (max=110, min=0). Higher scores indicate improvement. Lower scores indicate worsening. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint.
Time Frame: Baseline up to 2.5 years
Population: Full analysis set from combined studies.
Measure: Mean (95% Confidence Interval); unit: scores
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 921 | 909
scores
  Month 6 n=921,909 | 1.02 [0.46 to 1.59] | 0.64 [0.07 to 1.20]
  Month 12 n=879,863: number analyzed (Participants) | 879 | 863
  Month 12 n=879,863 | 1.82 [1.22 to 2.41] | 1.70 [1.10 to 2.30]
  Month 18 n=849,808: number analyzed (Participants) | 849 | 808
  Month 18 n=849,808 | 2.84 [2.24 to 3.45] | 2.05 [1.44 to 2.67]
  Month 24 n=492,468: number analyzed (Participants) | 492 | 468
  Month 24 n=492,468 | 3.50 [2.80 to 4.20] | 2.39 [1.67 to 3.11]
  Month 30 n=156,117: number analyzed (Participants) | 156 | 117
  Month 30 n=156,117 | 3.53 [2.39 to 4.68] | 2.97 [1.67 to 4.28]

19. Secondary Outcome: 6-month Confirmed Worsening of at Least 20% in the Timed 25-Foot Walk (T25FW) - Pooled Data
Description: The patient is directed to walk 25 feet quickly and safely as possible from one marked end to the other. The time is calculated from the initiation of the patient instructed to begin, until the patient has reached the 25-foot mark. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint.
Time Frame: Baseline, every 3 months up to 2.5 years
Population: Full analysis set from combined studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 936 | 925
percentage of participants
  Month 18 - from Kaplan Meier estimates | 11.0 [9.1 to 13.3] | 10.4 [8.5 to 12.6]
  Month 24 - from Kaplan Meier estimates | 11.4 [9.5 to 13.8] | 10.6 [8.7 to 12.9]

20. Secondary Outcome: 6-month Confirmed Worsening of at Least 20% in the 9-Hole Peg Test (9HPT) - Pooled Data
Description: 9-Hole Peg Test is a test of upper limb function. Participants place 9 pegs on pegboard and remove pegs and this is timed for each hand. Time recorded in seconds. Longer time indicates poorer upper limb function. 20% improvement is defined as 20% shorter time in seconds. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint.
Time Frame: Baseline, every 6 months up to 2.5 years
Population: Full analysis set from combined studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 932 | 920
percentage of participants
  Month 18 - from Kaplan Meier estimates | 2.9 [2.0 to 4.3] | 3.3 [2.3 to 4.8]
  Month 24 - from Kaplan Meier estimates | 2.9 [2.0 to 4.3] | 3.3 [2.3 to 4.8]

21. Secondary Outcome: 6-month Confirmed Disability Improvement (6mCDI) Sustained Until End of Study (EOS) as Measured by EDSS - Pooled Data
Description: A 6-month confirmed disability improvement (6mCDI) sustained until EOS was defined as a decrease from baseline EDSS sustained until EOS. For patients with a baseline EDSS of 0 to 1.5, no disability improvement was possible based on the protocol definition of an improvement; for patients with a baseline EDSS of ≥2 to 6 or ≥6.5 to 9.5, the criterion for disability improvement was a decrease in EDSS of ≤1 or ≤0.5, respectively. This study was not powered for the analysis of this endpoint individually. It was pre-specified in the study protocol to combine the data from this study with study COMB157G2301 to address this endpoint.
Time Frame: Baseline, every 3 months up to 2.5 years
Population: Full analysis set from combined studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 749 | 724
percentage of participants
  Month 18 - from Kaplan Meier estimates | 5.4 [4.0 to 7.4] | 4.6 [3.2 to 6.5]
  Month 24 - from Kaplan Meier estimates | 5.8 [4.2 to 7.8] | 4.6 [3.2 to 6.5]

22. Secondary Outcome: Number of New or Enlarging T2 Lesions on MRI Per Year From Month 12 Until End of Study (EOS)
Description: Number of new/enlarging T2 lesions on the last available MRI scan compared to Month 12 adjusted for different time of scans versus Month 12 due to variable follow up time in study.
Time Frame: Month 12 up to 2.5 years
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: T2 lesions per year
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 369 | 348
T2 lesions per year | 0.13 [0.09 to 0.18] | 3.84 [3.19 to 4.62]

23. Secondary Outcome: Percent Change in T2 Lesion Volume Relative to Baseline
Description: Percent change from baseline in total T2 lesion volume
Time Frame: Baseline, Month 12, Month 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage change in lesion volume
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 447 | 437
percentage change in lesion volume
  Month 12 n=447,437 | -2.4 (8.66) | 10.1 (38.57)
  Month 24 n=330,320: number analyzed (Participants) | 330 | 320
  Month 24 n=330,320 | -2.6 (9.34) | 17.8 (53.48)

24. Secondary Outcome: No Evidence of Disease Activity (NEDA-4)
Description: NEDA-4 was defined as no 3-month confirmed disability worsening, no confirmed MS relapse, no new or enlarging T2 lesions compared to baseline, and the annualized rate of brain atrophy >-0.04%.
Time Frame: Baseline, Month 12, Month 24
Population: Full analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 433 | 427
percentage of participants
  Month 12 n=433,427 | 23.8 [19.8 to 27.8] | 17.8 [14.2 to 21.4]
  Month 24 n=92,78: number analyzed (Participants) | 92 | 78
  Month 24 n=92,78 | 9.8 [3.7 to 15.9] | 5.1 [0.2 to 10.0]

25. Secondary Outcome: Multiple Sclerosis Impact Scale (MSIS-29) Physical Impact Score Change From Baseline
Description: MSIS-29 is a 29-item, self-administered questionnaire that includes 2 domains, physical and psychological. Responses are captured on a 4-point scale ranging from "not at all" (1) to "extremely" (4), where higher scores reflect greater impact on day to day life.
Time Frame: Baseline, every 6 months up to 2.5 years
Population: Full analysis set
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 473 | 461
scores on a scale
  Month 6 n=473,461 | -2.20 (0.652) | -0.46 (0.659)
  Month 12 n=448,438: number analyzed (Participants) | 448 | 438
  Month 12 n=448,438 | -2.47 (0.698) | -0.49 (0.704)
  Month 18 n=425,409: number analyzed (Participants) | 425 | 409
  Month 18 n=425,409 | -2.29 (0.784) | 1.53 (0.794)
  Month 24 n=235,238: number analyzed (Participants) | 235 | 238
  Month 24 n=235,238 | -2.93 (0.904) | 0.62 (0.905)
  Month 30 n=70,54: number analyzed (Participants) | 70 | 54
  Month 30 n=70,54 | -2.49 (1.270) | 1.44 (1.397)

26. Secondary Outcome: Multiple Sclerosis Impact Scale (MSIS-29) Psychological Impact Score Change From Baseline
Description: as for outcome 25
Time Frame: Baseline, every 6 months up to 2.5 years
Population: Full analysis set
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 473 | 461
scores on a scale
  Month 6 n=473,461 | -5.96 (0.807) | -3.77 (0.816)
  Month 12 n=448,436: number analyzed (Participants) | 448 | 436
  Month 12 n=448,436 | -5.42 (0.830) | -3.88 (0.839)
  Month 18 n=423,409: number analyzed (Participants) | 423 | 409
  Month 18 n=423,409 | -6.23 (0.884) | -2.51 (0.896)
  Month 24 n=234,238: number analyzed (Participants) | 234 | 238
  Month 24 n=234,238 | -6.10 (1.092) | -3.12 (1.090)
  Month 30 n=70,54: number analyzed (Participants) | 70 | 54
  Month 30 n=70,54 | -6.25 (1.623) | -4.75 (1.797)

27. Secondary Outcome: Annualized Relapse Rates (ARR) by NfL High-low Subgroups - Pooled Data
Description: ARR was the number of confirmed relapses in a year, calculated as the total number of relapses for all participants in the treatment group divided by the total participant-years of time in study. A confirmed MS relapse was defined as one accompanied by a clinically-relevant change in the EDSS performed by the Independent EDSS rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores or 2 points on one functional score (excluding changes involving bowel/bladder or cerebral functional system).
Time Frame: Baseline up to 2.5 years
Population: Supportive sub-group analysis based on estimations from pooled data from this study and study COMB157G2301.
Measure: Mean (95% Confidence Interval); unit: number of relapses in a year
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 871 | 841
number of relapses in a year
  High > median n=443,410: number analyzed (Participants) | 443 | 410
  High > median n=443,410 | 0.08 [0.07 to 0.11] | 0.21 [0.17 to 0.26]
  Low <= median n=428,431: number analyzed (Participants) | 428 | 431
  Low <= median n=428,431 | 0.12 [0.09 to 0.15] | 0.23 [0.19 to 0.27]

28. Secondary Outcome: Number of New or Enlarging T2 Lesions Per Year by NfL High-low Subgroups - Pooled Data
Description: Number of new or enlarging T2 lesions on MRI per year (annualized lesion rate).
Time Frame: Baseline, yearly up to 2.5 years
Population: Supportive sub-group analysis based on estimations from pooled data from this study and study COMB157G2301.
Measure: Mean (95% Confidence Interval); unit: T2 lesions per year
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 850 | 823
T2 lesions per year
  High > median n=432,402: number analyzed (Participants) | 432 | 402
  High > median n=432,402 | 0.95 [0.82 to 1.11] | 5.28 [4.61 to 6.03]
  Low <= median n=418,421: number analyzed (Participants) | 418 | 421
  Low <= median n=418,421 | 0.39 [0.33 to 0.47] | 3.02 [2.64 to 3.46]

29. Secondary Outcome: Brain Volume Loss by NfL High-low Subgroups - Pooled Data
Description: as for outcome 11
Time Frame: Baseline, Months 12 and 24
Population: Supportive sub-group analysis based on estimations from pooled data from this study and study COMB157G2301.
Measure: Mean (95% Confidence Interval); unit: percentage of brain volume loss
Arm/Group | OMB 20 mg | TER 14 mg
Number analyzed (Participants) | 819 | 794
percentage of brain volume loss
  High > median n=416,387: number analyzed (Participants) | 416 | 387
  High > median n=416,387 | -0.32 [-0.38 to -0.26] | -0.43 [-0.49 to -0.37]
  Low <= median n=403,407: number analyzed (Participants) | 403 | 407
  Low <= median n=403,407 | -0.24 [-0.30 to -0.18] | -0.29 [-0.35 to -0.22]

30. Secondary Outcome: Pharmacokinetic (PK) Concentrations of Ofatumumab
Description: Summary statistics of pharmacokinetic (PK) concentrations from trough samples collected within a 7-day window prior or at day of dosing.
Time Frame: Baseline, Weeks 4, 12, 24, 48, 96
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | OMB 20 mg
Number analyzed (Participants) | 481
ug/mL
  Baseline n=325: number analyzed (Participants) | 325
  Baseline n=325 | 0.00325 (0.031372)
  Week 4 n=346: number analyzed (Participants) | 346
  Week 4 n=346 | 1.26512 (0.964645)
  Week 12 n=257: number analyzed (Participants) | 257
  Week 12 n=257 | 0.20932 (0.287839)
  Week 24 n=243: number analyzed (Participants) | 243
  Week 24 n=243 | 0.38203 (0.433175)
  Week 48 n=240: number analyzed (Participants) | 240
  Week 48 n=240 | 0.59087 (0.594490)
  Week 96 n=304: number analyzed (Participants) | 304
  Week 96 n=304 | 1.13218 (0.991141)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until last administration of study treatment plus 100 days post treatment, up to maximum duration of approximately 2.7 years
Groups:
- OMB 20mg: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter (+ teriflunomide-matching placebo capsule orally once daily)
- TER 14mg: Teriflunomide 14 mg capsule orally once daily (+ ofatumumab-matching placebo injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter)
Arm/Group | OMB 20mg | TER 14mg
All-Cause Mortality (participants affected / at risk) | 0/481 | 1/474
Serious Adverse Events (participants affected / at risk) | 42/481 | 37/474
Other Adverse Events (participants affected / at risk) | 348/481 | 322/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OMB 20mg (N=481) | TER 14mg (N=474)
Bundle branch block bilateral (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 5 | 1
Cystitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Headache (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Quadriplegia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Testicular infarction (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 2
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Bundle branch block bilateral (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 5 | 1
Cystitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Headache (Nervous system disorders) | 2 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 1 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Quadriparesis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Testicular infarction (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 2
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OMB 20mg (N=481) | TER 14mg (N=474)
Diarrhoea (Gastrointestinal disorders) | 28 | 49
Nausea (Gastrointestinal disorders) | 30 | 32
Fatigue (General disorders) | 25 | 32
Injection site reaction (General disorders) | 61 | 26
Influenza (Infections and infestations) | 30 | 30
Nasopharyngitis (Infections and infestations) | 88 | 87
Upper respiratory tract infection (Infections and infestations) | 49 | 47
Urinary tract infection (Infections and infestations) | 54 | 35
Injection related reaction (Injury, poisoning and procedural complications) | 119 | 66
Blood immunoglobulin M decreased (Investigations) | 30 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 30
Headache (Nervous system disorders) | 68 | 65
Anxiety (Psychiatric disorders) | 28 | 17
Depression (Psychiatric disorders) | 24 | 24
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 74
Hypertension (Vascular disorders) | 20 | 31
Diarrhoea (Gastrointestinal disorders) | 28 | 49
Nausea (Gastrointestinal disorders) | 30 | 32
Fatigue (General disorders) | 25 | 32
Injection site reaction (General disorders) | 61 | 26
Influenza (Infections and infestations) | 27 | 28
Nasopharyngitis (Infections and infestations) | 88 | 88
Upper respiratory tract infection (Infections and infestations) | 52 | 47
Urinary tract infection (Infections and infestations) | 55 | 34
Injection related reaction (Injury, poisoning and procedural complications) | 119 | 66
Blood immunoglobulin M decreased (Investigations) | 31 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 30
Headache (Nervous system disorders) | 69 | 66
Anxiety (Psychiatric disorders) | 30 | 17
Depression (Psychiatric disorders) | 23 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 24
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 75
Hypertension (Vascular disorders) | 20 | 32

LIMITATIONS AND CAVEATS:
This study was not powered for the analysis of some secondary endpoints as a stand-alone study. It was pre-specified in the study protocol to combine the data with study COMB157G2301 to address these endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT02792231/Prot_001.pdf
  • Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT02792231/SAP_000.pdf